CLINICAL TRIAL: NCT07349394
Title: A Phase 1, Open-label, Drug-Drug Interaction Study to Evaluate the Effect of Multiple Doses of Vanzacaftor/Tezacaftor/Deutivacaftor on the Pharmacokinetics of Rosuvastatin in Healthy Subjects
Brief Title: Effect of Vanzacaftor/Tezacaftor/Deutivacaftor (VNZ/TEZ/D-IVA) on the PK of Rosuvastatin in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX25-121-014
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — deutivacaftor, tezacaftor , vanzacaftor; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VNZ/TEZ/D-IVA and Rosuvastatin (Experimental): Rosuvastatin will be administered to participants as a single oral dose on Day 1 and then co-administered with VNZ/TEZ/D-IVA on Day 18.VNZ/TEZ/D-IVA dose will be administered once daily (qd) from Day 5 to Day 22.
  Interventions: Drug: VNZ/TEZ/D-IVA; Drug: Rosuvastatin

INTERVENTIONS:
Drug: VNZ/TEZ/D-IVA — Fixed-dose combination (FDC) Tablet for oral administration.
  Other Names: Vanzacaftor/Tezacaftor/Deutivacaftor; VX-121/VX-661/VX-561; VX-121/VX-661/CTP-656
Drug: Rosuvastatin — Tablet for oral administration.

SUMMARY:
The purpose of this study is to evaluate the effect of multiple doses of vanzacaftor/tezacaftor/deutivacaftor (VNZ/TEZ/D-IVA) on the PK of rosuvastatin and the safety and tolerability of coadministration of VNZ/TEZ/D-IVA with rosuvastatin.

DETAILED DESCRIPTION:
The study is being conducted to evaluate the effect of multiple doses of VNZ/TEZ/D-IVA on the PK of rosuvastatin and the safety and tolerability of coadministration of VNZ/TEZ/D-IVA with rosuvastatin in healthy participants.

Note: This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR11.60and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24and11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2), both inclusive
* A total body weight greater than (>)50 kg

Key Exclusion Criteria:

* History of febrile illness within 5 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Female participants who are pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last dose of the study drug
* Male participants with a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last dose of the study drug

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Rosuvastatin in the Absence and Presence of VNZ/TEZ/D-IVA | Day 1 up to Day 23
Area Under the Concentration Time-curve (AUC) of Rosuvastatin in the Absence and Presence of VNZ/TEZ/D-IVA | Day 1 up to Day 23

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 39

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences - Kansas City, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/